CLINICAL TRIAL: NCT05354219
Title: Validation and Reliability of Iris Recognition and Manual InfraRed Cameras Using Bespoke Image Analysis Software for the Quantification of Corneal Opacification in Mucopolysaccharidoses
Brief Title: Validation and Reliability of Iris Cameras in Mucopolysaccharidoses
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Manchester University NHS Foundation Trust (Other Government)
Collaborators: Orchard Therapeutics (Industry)
Responsible Party: Sponsor
Other Study IDs: IRAS 315339
Record Dates: First submitted 2022-04-12; First posted 2022-04-29 (Actual); Last update posted 2023-03-22 (Actual); Status verified 2023-03

CONDITIONS: Mucopolysaccharidoses
MeSH Terms: conditions — Mucopolysaccharidoses | interventions — X-Rays

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- MPS patients: Any patient aged 0-100 with MPS type I, type III, type IV and type VI. Type VII MPS patients may also be eligible.
  Interventions: Other: Imaging
- Control: For the control group -
  Participants of any age currently being followed at MREH that have an eye condition unrelated to the cornea as established by clinical examination.
  Interventions: Other: Imaging

INTERVENTIONS:
Other: Imaging — Imaging with 3 iris cameras

SUMMARY:
To assess the reliablity and validity of 2 new iris cameras in the assement of corneal opacification in mucopolysaccharidoses

DETAILED DESCRIPTION:
The mucopolysaccharidoses (MPS) are a group of disorders resulting from accumulation of glycosaminoglycans within various tissues including the eye. This can result in visual loss from corneal opacification. The assessment of corneal opacification is extremely subjective and based on a clinician grading this during slit lamp examination. There can be a significant variability and can prove problematic particularly in clinical trials assessing if corneal opacification is affected by potential new treatments.

The use of imaging could facilitate objective measurement of corneal clouding. A previous study using an iris camera and image analysis to provide a corneal opacification measure score (COM score) demonstrated that it can be used in children with MPS, however it still had limitations- as the system is fully automated, if certain conditions are not met an image is not captured. This can be an issue in younger children who may not be cooperative, and limited its use in younger patient populations.

It is anticipated that these limitations can be addressed by employing a newer iris camera (IriShield MK2120UL). The new camera's advantage is that it takes images monocularly, therefore only the eye under question needs to be aligned. We will also assess a new manual system (IRcamNew) which takes images whenever the shutter is manually pressed. This would be useful in children who cannot fixate with one eye, and can also be used when the child is examined under general anaesthetic which is commonly done in paediatric ophthalmology.

If proven to be comparable to the existing iris camera (IriscamOrig) in terms of validity and reliability, the added benefits of these new iris cameras can open its use in a wider range of patient populations - for instance, in paediatric clinical trials-, as well as allowing longitudinal tracking of corneal clouding from early childhood well into adulthood.

ELIGIBILITY:
Inclusion Criteria:

* Any patient aged 0-100 with MPS type I, type III, type IV and type VI. Type VII MPS patients may also be eligible.

For the control group -

Participants of any age currently being followed at MREH that have an eye condition unrelated to the cornea as established by clinical examination.

Exclusion Criteria:

* MPS II

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: MPS patients and healthy controls
Sampling Method: Non-Probability Sample
Enrollment: 60 (Estimated)
Dates: Start 2023-03-08 (Actual); Primary Completion 2023-09-08 (Estimated); Study Completion 2023-09-08 (Estimated)

PRIMARY OUTCOMES:
Comparison of reliability of images taken by two different operators using the two ne w iris cameras | 2 months
  Bland altman plots to compare reliability between images and COM scores obtained by 2 different operators
Correlation of COM scores between two new iris cameras and IrisCamOrig | 2 months
  Validity will be assessed by comparing the COM scores generated by the new iris cams to the previously validated iris camera

SECONDARY OUTCOMES:
Comparison of clinical grading to COM score obtained by image analysis | 1 month
  Compare clinical grading of corneal opacification on slit lamp by clinicians to corneal opacification measure generated by image analysis

CONTACTS AND LOCATIONS:
Locations (1):
- Manchester University NHS Foundation Trust, Manchester, United Kingdom

IPD SHARING:
Plan to Share IPD: Undecided